CLINICAL TRIAL: NCT03025438
Title: Cytological Diagnosis of Hepatic Angiosarcoma and Its Histopathologic Correlation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201603013RINA
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-01

CONDITIONS: Hepatic Angiosarcoma
Keywords: angiosarcoma; Cytology; liver; cancer
MeSH Terms: conditions — Hemangiosarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cytological diagnosis of hepatic angiosarcoma by fine-needle aspiration (FNA) or imprint cytology is difficult due not only to its various cytomorphologic features but also clinical rarity. Vasoformative features, such as pseudo-acini, branching pseudo-capillary structure, and intracytoplasmic lumina, are clues to achieve the diagnosis. But these features are not always present. In order to find clues for cytological diagnosis of angiosarcoma, we collected cases of hepatic angiosarcoma to study their cytological features. And then compared these features with those in their histopathological biopsy or resection.

DETAILED DESCRIPTION:
Hepatic angiosarcoma is a rare hepatic malignant tumor. Although diagnosis of hepatic angiosarcoma by FNA cytology has been reported since 1982, followed by several studies, its cytomorphologic features were still not well recognized by cytopathologists because of its clinical rarity and various morphologic features.

We reviewed literatures about cytomorphology of hepatic angiosarcoma by FNA. There are only 11 cases retrieved in 10 articles searched from Medline. The sex M/F ratio was 6/4 (one unknown); age range was 56 to 79 years old. In initial cytological evaluation, four cases got angiosarcoma or consistent/suspicious angiosarcoma diagnosis. Positive for malignancy, sarcoma, and poorly differentiated spindle cell lesion were in one case respectively. One was diagnosed as atypical cells. Remaining three were unavailable by their reports.

In cytological morphologic features, all but one met least 2 of 3 cytological cellular criteria of angiosarcoma cells: spindle cells, epithelioid cells, and pleomorphic cells. In cytological architectural features, 7 of 11 cases showed vasoformative structures; 5 of 11 cases showed intracytoplasmic lumen or erythrophagocytosis. Ten of 11 cases had histologic/pathologic confirmation as angiosarcoma. One case reported interrelation of tumor structures and their own accompanied liver tissue in cell blocks.

ELIGIBILITY:
Inclusion criteria:

Consecutive patients of hepatic angiosarcoma performed FNA and/or imprint cytological examinations in our hospital.

Exclusion criteria:

1. Patients without pathological confirmation.
2. Patients who are not angiosarcoma by pathological reviews.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of a medical center in Taiwan; National Taiwan University Hospital (NTUH)
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-02-04 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
all cause mortality | about 10 years from the date of diagnosis to the last follow-up date by medical record

CONTACTS AND LOCATIONS:
Overall Officials: Wern-Cherng Cheng, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Department of laboratory medicine, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided